CLINICAL TRIAL: NCT05198596
Title: A Phase III, Parallel Group, Prospective, Randomized, Double-blind, Active-controlled, Two-arm, Multi-center Study to Evaluate the Immunogenicity, Safety, and Tolerability of MVC-COV1901 Compared to AZD1222 in Adult of 18 Years and Above
Brief Title: A Study to Evaluate Immunogenicity and Safety of MVC-COV1901 Compared With AZD1222 in Adults Aged 18 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT-COV-32
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Vaccine
Keywords: COVID-19 Vaccine
MeSH Terms: interventions — MVC-COV1901 vaccine; ChAdOx1 nCoV-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVC-COV1901 (Experimental): S-2P protein with CpG and Aluminum Hydroxide/0.5mL
  Interventions: Biological: MVC-COV1901
- AZD1222 (Active Comparator): ChAdOx1 nCoV-19 vaccine
  Interventions: Biological: AZD1222

INTERVENTIONS:
Biological: MVC-COV1901 — Approximately125 participants will receive 2 doses of MVC-COV1901(S-2P protein with adjuvant) at Day 1 and Day 29 via intramuscular (IM) injection in the deltoid region
  Arms: MVC-COV1901
Biological: AZD1222 — Approximately 125 participants will receive 2 doses of AZD1222 at Day 1 and Day 29 via intramuscular (IM) injection in the deltoid region
  Arms: AZD1222

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of MVC- COV1901 vaccine compared to AZD1222 in heathy adults.

DETAILED DESCRIPTION:
The primary objective of the study is to measure the anti-SARS-CoV-2 neutralizing antibody titres in adult participants so as to demonstrate immunogenic superiority of MVC-COV1901 to the active control, AZD1222 vaccine, in terms of the GMT of neutralizing antibodies at 14 days after the second dose of the study intervention. This study also assesses the safety and tolerability of the study intervention and explores the immunogenicity in terms of antigen-specific immunoglobulin as well as the potential efficacy of MVC-COV1901 in preventing COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged 18 years and above at randomization.
2. Healthy adult or adult with pre-existing medical conditions who is in a stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease 3 months before enrollment and expected to remain stable for the duration of the study.
3. Female participant:

   1. A female participant is eligible if the participant is a woman of non-childbearing potential, i.e., surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal.
   2. If the participant is a woman of childbearing potential, she must agree to practice sexual abstinence or agree to use medically effective contraception from 14 days before screening to 30 days following the last administration of study intervention. Highly effective methods of contraception include:

   i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine hormonal-releasing system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository iii. Azoospermic partner (vasectomized or due to medical cause), provided the partner is the sole sexual partner of the female participant and the absence of sperm has been confirmed (from medical records/examination/history).

   c.Have a negative pregnancy test
4. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
5. Participant or the participant's legal representative must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding or have plan to become pregnant within 30 days after the last administration of the study intervention.
2. Employees at the investigator's site, of the Sponsor or delegate (e.g., contract research organization) who are directly involved in the conduct of the study.
3. Currently receiving or received any investigational intervention within 30 days prior to the first dose of the study intervention.
4. Administered any licensed live-attenuated vaccines within 28 days or other licensed non- live-attenuated vaccines within 7 days prior to the first dose of the study intervention.
5. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the first dose of the study intervention.
6. Currently receiving or anticipate receiving concomitant immunosuppressive or immune- modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the first dose of the study intervention.
7. Currently receiving or anticipate receiving treatment with tumor necrosis factor (TNF)-α inhibitors, e.g., infliximab, adalimumab, etanercept within 12 weeks prior to the first dose of the study intervention.
8. Major surgery or any radiation therapy within 12 weeks prior to the first dose of the study intervention.
9. Has received any other investigational or approved COVID-19 vaccine.
10. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
11. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
12. Bleeding disorder considered a contraindication to intramuscular (IM) injection or phlebotomy.
13. Documented SARS-CoV-2 infection prior to the first dose of study intervention, or an individual with positive anti-SARS-CoV-2 antibody test at screening (including rapid tests).
14. A history of cerebral venous sinus thrombosis, heparin-induced thrombocytopenia, thrombosis with thrombocytopenia syndrome (TTS), antiphospholipid syndrome, or capillary leak syndrome.
15. Participant who, in the investigator's judgement, is not in a stable condition and by participating in the study could adversely affect the safety of the participant, interfere with adherence to study requirements or evaluation of any study endpoint. This may include a participant with ongoing acute diseases, severe infections, autoimmune disease, laboratory abnormality or serious medical conditions in the following systems: cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, or psychiatric.
16. A history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901 or AZD1222.
17. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of neutralizing antibody (GMT) | Day 1 to Day 43
  To demonstrate the immunogenic superiority of MVC-COV1901 to AZD1222 in terms of neutralizing antibody titers at 14 days after the second vaccination
  -GMT ratio
Incidence of Adverse Event within 28 days post the second study intervention | Day 1 to Day 57
  To evaluate the safety and tolerability of MVC-COV1901 compared to AZD1222 from Day 1 to 28 days after the second vaccination
  The number and percentage of participants with the occurrence of:
  * Solicited local AEs
  * Solicited systemic AEs
  * Unsolicited AEs
  * Medically attended AEs (MAAEs) • AESIs
  * VAED
  * SAEs

SECONDARY OUTCOMES:
Immunogenicity of neutralizing antibody (GMT) | Day 29 to Day 209
  To evaluate the immunogenicity of MVC-COV1901 compared to AZD1222 in terms of neutralizing antibody titers from Day 29 to Day 209
  • GMT
Immunogenicity of neutralizing antibody(SCR) | Day 29 to Day 209
  To evaluate the immunogenicity of MVC-COV1901 compared to AZD1222 in terms of neutralizing antibody titers from Day 29 to Day 209
  • SCR
Immunogenicity of neutralizing antibody(GMT ratio) | Day 29 to Day 209
  To evaluate the immunogenicity of MVC-COV1901 compared to AZD1222 in terms of neutralizing antibody titers from Day 29 to Day 209
  • GMT ratio
Incidence of Adverse Event throughout study conduct | Day 1 to Day 209
  To evaluate the safety of MVC COV1901 compared to AZD1222 over the study period
  The number and percentage of participants with the occurrence of:
  * MAAEs
  * AESIs
  * VAED
  * SAEs

OTHER OUTCOMES:
Incidence of confirmed COVID-19 cases | Day 15 to Day 209
  To estimate the efficacy of MVC-COV1901, as compared to AZD1222, in the prevention of COVID-19 in terms of :
  * The number of laboratory-confirmed COVID-19 cases occurring ≥ 15 days after any dose of study intervention.
  * The number of laboratory-confirmed COVID-19 severe cases occurring ≥ 15 days after any dose of study intervention.
Immunogenicity of antigen-specific immunoglobulin titers(GMT) | Day 29 to Day 209
  To evaluate the immunogenicity of MVC-COV1901 compared to AZD1222 in terms of antigen-specific immunoglobulin titers from Day 29 to Day 209
  • GMT
Immunogenicity of antigen-specific immunoglobulin titers(SCR) | Day 29 to Day 209
  o evaluate the immunogenicity of MVC-COV1901 compared to AZD1222 in terms of antigen-specific immunoglobulin titers from Day 29 to Day 209
  • SCR
Immunogenicity of antigen-specific immunoglobulin titers(GMT ratio) | Day 29 to Day 209
  To evaluate the immunogenicity of MVC-COV1901 compared to AZD1222 in terms of antigen-specific immunoglobulin titers from Day 29 to Day 209
  • GMT ratio
Cell Mediated Immunity | Day 1 to Day 43
  To assess cell-mediated immune response of MVC-COV1901compared to AZD1222

CONTACTS AND LOCATIONS:
Overall Officials: Allen Lien, MD. Dr.PH, Study Director — Medigen Vaccine Biologics
Locations (2):
- Thailand (2):
  - College of Medicine and Public Health, Ubon Ratchathani University, Warin Chamrap, Changwat Ubon Ratchathani
  - Sunpasitthiprasong Hospital, Ubon Ratchathani